CLINICAL TRIAL: NCT01908335
Title: Phase Ⅱ, Multi-center, Randomized, Open-label, Parallel-group, Active Controlled Study for the Efficacy and Safety of Pegylated Recombinant Consensus Interferon Variant Solution for Injection in the Treatment of Chronic Hepatitis C
Brief Title: A Phase Ⅱ Dose-escalating Study of PEG-IFN-SA and Ribavirin in IFN Naive Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Kawin Technology Share-Holding Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Cheng jun, vice president, Beijing Kawin Technology Share-Holding Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAWIN-002-1
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Hepatitis C
Keywords: interferon; ribavirin; virological response
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — PEG-IFN-SA; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (PEG-IFN-SA /RBV low dose) (Experimental): PEG-IFN-SA 0.75μg/kg/week and RBV 1000mg-1200mg/d bid depending on body weight(BW),（BW<75kg，1000mg/d；BW≥75kg，1200mg/d）
  Interventions: Drug: PEG-IFN-SA /RBV low dose
- B (PEG-IFN-SA /RBV middle dose) (Experimental): PEG-IFN-SA 1.5μg/kg/week and RBV 1000mg-1200mg/d bid depending on body weight(BW),（BW<75kg，1000mg/d；BW≥75kg，1200mg/d）
  Interventions: Drug: PEG-IFN-SA /RBV middle dose
- C (PEG-IFN-SA /RBV high dose) (Experimental): PEG-IFN-SA 2.0μg/kg/week and RBV 1000mg-1200mg/d bid depending on body weight(BW),（BW<75kg，1000mg/d；BW≥75kg，1200mg/d）
  Interventions: Drug: PEG-IFN-SA /RBV high dose
- D (Pegasys /RBV) (Active Comparator): Pegasys 180μg/week and RBV 1000mg-1200mg/d bid depending on body weight(BW),（BW<75kg，1000mg/d；BW≥75kg，1200mg/d）
  Interventions: Drug: Pegasys /RBV

INTERVENTIONS:
Drug: PEG-IFN-SA /RBV low dose — 24 weeks for genotype 2,3 and 48 weeks for non-genotype2,3
  Arms: A (PEG-IFN-SA /RBV low dose)
Drug: PEG-IFN-SA /RBV middle dose — 24 weeks for genotype 2,3 and 48 weeks for non-genotype2,3
  Arms: B (PEG-IFN-SA /RBV middle dose)
Drug: PEG-IFN-SA /RBV high dose — 24 weeks for genotype 2,3 and 48 weeks for non-genotype2,3
  Arms: C (PEG-IFN-SA /RBV high dose)
Drug: Pegasys /RBV — 24 weeks for genotype 2,3 and 48 weeks for non-genotype2,3
  Arms: D (Pegasys /RBV)

SUMMARY:
This dose-escalating study is to evaluate the efficacy and the safety of different doses of a new bio-product Pegylated Recombinant Consensus Interferon Variant Solution for Injection (PEG-IFN-SA) and Ribavirin（RBV） in the treatment of Chronic hepatitis C who have not been previously treated with Interferon(IFN) by exploring the dose-effect relationship, while identity the optimal dose for phase Ⅲ study. In addition, population pharmacokinetic method is adopted to assess the pharmacokinetic behavior, individuals / intra-individual variability, and the possible factors for further study.

DETAILED DESCRIPTION:
Total 200 subjects will be randomized and enrolled into four groups proportionally receiving experimental drug of high dose, middle dose, low dose and positive-control drug. Treatment duration will be 24 or 48 weeks corresponding to different HCV genotype, genotype 2,3 and non-genotype2,3.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65 years
* Body Mass Index (BMI) 18-30
* Chronic hepatitis C , diagnosed according to Chinese guideline of Hepatitis C (year 2004)
* Detectable serum HCV-RNA by quantitative polymerase chain reaction assay and positive anti-HCV antibody
* Female subjects of childbearing age with no history of menopause and negative pregnancy test, both female and male( including their partners ) subjects were required to conduct adequate contraception since screening until the 6 months after treatment
* Volunteered to participate in this study, understood and signed an informed consent

Exclusion Criteria:

* Previous IFN treated patients
* Co-infection with HAV, HBV, HEV, EBV, CMV and HIV
* Evidences of hepatic decompensation, including but not limited to serum total bilirubin> 2 times the upper limit of normal (ULN); serum albumin <35g/L; prothrombin activity (PTA) <60%; ascites, upper gastrointestinal bleeding and hepatic encephalopathy; Child-Pugh score B/C grade
* Hepatotoxic drugs was used for a long time within past 6 months
* Diagnosed with primary hepatocellular carcinoma or supported by evidences including but not limited to AFP> l00ng/ml, suspicious liver nodules by imaging examinations
* Liver diseases from causes other than HCV infection, including alcoholic liver disease, non-alcoholic steatohepatitis, drug-induced hepatitis, autoimmune hepatitis (antinuclear antibody titer higher than 1:100), hepatolenticular degeneration (Wilson's disease) and hemochromatosis, etc.
* White blood cell count <3×109/L; Neutrophil count<1.5×109/L; platelet count<90×109/L; hemoglobin below the lower limit of normal
* Serum creatinine not within the normal range
* Serum creatine kinase> 3 ULN
* Positive thyroid antibodies (A-TPO, A-TG)
* Therapy with potent immunomodulatory agents such as adrenocorticotropic hormone, thymosin α1 etc. within past 6 months or an anticipated usage during the period of study
* Allergies or severe allergies, especially allergic to study drugs or any ingredients of the study drugs
* Severe autoimmune diseases; psychiatric and nervous system disorders, including history of Psychiatric illness or with family history (especially depression, depressive tendencies, epilepsy and hysteria, etc.); Serious blood disorders (all kinds of anemia, hemophilia, etc.); Severe kidney disease (chronic kidney disease, renal insufficiency, etc.); poorly controlled digestive diseases; endocrine disorders such as thyroid disease and diabetes; severe respiratory disease (pneumonia, chronic obstructive pulmonary disease, interstitial lung disease, etc.); cardiovascular diseases (hypertension, uncontrolled coronary atherosclerotic heart disease, heart failure, etc.); retinal disease; malignancies; or unsuitable for study considered by clinician
* Function organs transplant
* Evidence of alcohol or drug abuse (average alcohol consumption male> 40g / day, female> 20g / day)
* Pregnant or lactating women
* Usage of prohibition drugs in this study
* Participated in other clinical trials 3 months prior to the screening
* Unwilling to sign the informed consent and adhere to treatment requirements
* Other conditions not suitable for study judged by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
cEVR (complete early virologic response) | weeks 12 of study therapy
  defined as the proportion of patients who had undetectable plasma HCV RNA at weeks 12

SECONDARY OUTCOMES:
Proportion of patients who had undetectable plasma HCV RNA | weeks 4, 24, 48 of study therapy and 24 weeks after the end of treatment
HCV RNA load reduction | weeks 4, 12, 24, 48 of study therapy and 24 weeks after the end of treatment
eRVR ( extended rapid virologic response) | weeks 4 and 12 of study therapy
  defined as the proportion of patients who had undetectable plasma HCV RNA at weeks 4 and 12
Breakthrough | weeks 24, 48 of study therapy
  defined as the proportion of patients who had detectable plasma HCV RNA at any point during treatment after virological response( undetectable plasma HCV RNA)
Relapse | 12 and 24 weeks after the end of treatment
  defined as the proportion of patients who had undetectable HCV RNA at the end of treatment, but reappearance of HCV RNA after then

CONTACTS AND LOCATIONS:
Overall Officials: Cheng jun, MD, PhD, Principal Investigator — Beijing Ditan Hospital
Locations (52):
- China (52):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical Unbiversity, Guangzhou, Guangdong
  - The third people's hospital of Shenzhen, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Third Affiliated Hospital, Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College Huazhong University of Science ＆ Technology, Wuhan, Hubei
  - Union hospital, Tongji Medical College Huazhong University of Science ＆ Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - Jiangsu province hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - The first affiliated hospital of suzhou university, Suzhou, Jiangsu
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital (Yanbian Hospital), Yanji, Jilin
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - First Affiliated Hospital Of Medical College of Xian Jiaotong University, Xi'an, Shaanxi
  - Second Affiliated Hospital Of Medical College of Xian Jiaotong University, Xi'an, Shaanxi
  - Tangdu Hospital , , Fourth Military Medical University, Xi'an, Shaanxi
  - Jinan Infectious Disease Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong university, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Academy of Medical Science ＆Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Xixi Hospital of Hangzhou, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - 302 Military Hospital of China, Beijing
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Beijing Youyi Hospital, capital Medical University, Beijing
  - General Hospital of Beijing Military Region, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Chongqing Southwest Hospital, Chongqing
  - Daping Hospital, Research Institute of Surgery Third Military Medical University, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Ruijing Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Tianjin Infectious Disease Hospital, Tianjin